CLINICAL TRIAL: NCT06830954
Title: Bioequivalence Study of Fluvastatin Sodium Extended Release Tablets in Healthy Participants
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shenzhen Salubris Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SAL-138-BE01
Record Dates: First submitted 2025-02-10; First posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Bioequivalence
Keywords: Fluvastatin; Pharmacokinetics; Bioequivalence

STUDY DESIGN:
Intervention Model Description: two-sequence, four-period
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Drug: Fluvastatin sodium extended release tablet, 80 mg The participants randomly received single oral dose of Fluvastatin sodium extended release tablet 80 mg.
  Interventions: Drug: Group A; Drug: Reference Group
- Group B (Active Comparator): Drug: Fluvastatin sodium extended release tablet, 80 mg The participants randomly received single oral dose of Fluvastatin sodium extended release tablet 80 mg.
  Interventions: Drug: Group A; Drug: Reference Group

INTERVENTIONS:
Drug: Group A — Drug: Fluvastatin sodium extended release tablet, 80 mg Period 1 and 3, the participants randomly received single oral dose of test drug ( Fluvastatin sodium extended release tablet 80 mg). Period 2 and 4, the participants randomly received single oral dose of reference drug ( Fluvastatin sodium extended release tablet 80 mg).
  Other Names: Test Group
Drug: Reference Group — Drug: Fluvastatin sodium extended release tablet, 80 mg Period 1 and 3, the participants randomly received single oral dose of reference drug ( Fluvastatin sodium extended release tablet 80 mg). Period 2 and 4, the participants randomly received single oral dose of test drug ( Fluvastatin sodium extended release tablet 80 mg).

SUMMARY:
The purpose of this study is to evaluate the bioequivalence of the test preparation (Fluvastatin sodium extended release tablet, 80 mg) manufactured by Shenzhen Salubris Pharmaceuticals Co., Ltd. and the reference preparation (80 mg) manufactured by Beijing Novartis Pharma Co., Ltd. in healthy participants under fasting and fed conditions.

DETAILED DESCRIPTION:
This is a single center, open-label, randomized, two-sequence, four-period, crossover bioequivalence study.

The study is mainly divided into two stages: screening period (2 weeks) and treatment period (4 weeks). Washout time is 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Participants have fully understood the trial's objectives, procedures, and potential adverse effects, and voluntarily signed informed consent form prior to the trial.
* Participants are able to communicate effectively with the investigator and comply with the protocol requirements to complete the trial.
* Healthy male or female adults aged 18 to 65 years (inclusive).
* Body weight ≥50 kg for male participants and ≥45 kg for female participants at screening, with a body mass index (BMI) between 19.0 and 26.0 kg/m2 (inclusive; BMI = body weight ÷ height2).
* No abnormalities or only slight abnormalities not clinically significant of tests/examinations as judged by the investigator. Alanine aminotransferase (ALT), aspartate aminotransferase (AST), and creatine kinase (CK) must not exceed the upper limit of the normal reference range.

Participants or their partners must not have any pregnancy plans during the study and for three months after the last administration of the investigational drug. They must voluntarily take effective contraceptive measures (the use of contraceptive medications is prohibited during the study) to avoid pregnancy for themselves or their partners, and participants must not donate sperm or eggs (ovum and oocytes) for reproductive or assisted reproductive purposes.

Exclusion Criteria:

* Pregnant or lactating women, or women of child-bearing potential (WOCBP) with a positive pregnancy test at screening.
* Participants who have a history of clinically significant acute allergy to drug or food within two weeks prior to screening, or have an allergic constitution (e.g., allergy to two or more drugs, food, or pollens), or have a history of allergic diseases (e.g., asthma, urticaria, eczematous dermatitis, etc.), or have possible or definite allergy, hypersensitivity or clinically significant reactions to investigational drugs or excipients judged by the investigator.
* Participants with any disease (e.g., acute gastritis, peptic ulcer, anaphylactoid purpura, lupus erythematosus, etc.) or history (e.g., haemorrhage intracranial, hemorrhage intraocular, haemophilia, angiohaemophilia, etc.) that may change or aggravate haemorrhagic diathesis as judged by the investigator.
* Participants with a positive result for any of the following tests: hepatitis B surface antigen test, hepatitis C antibody test, HIV antibody test, and treponema pallidum antibody test.
* Drug abuse, alcohol abuse, or tobacco addiction:

Participants with a history of drug abuse, or a positive result for drug abuse test at screening; Participants with an average alcohol consumption of more than 14 units per week (1 unit ≈ 17.7 mL of ethanol, i.e., 1 unit ≈ 360 mL of beer with 5% alcohol content or 45 mL of spirit with 40% alcohol content or 150 mL of wine with 12% alcohol content) within 3 months prior to screening, or with a positive result for breath alcohol test at screening, or those who could not completely stop consuming alcohol-containing food or beverages during the study; Participants with an average tobacco consumption of more than 5 cigarettes per day within 3 months prior to screening, or those who could not completely stop consuming tobacco products during the study.

•Subjects who used any of the following food, medications, or treatments prior to the first dose: Used any drugs that inhibit or induce liver drug metabolism (e.g., inducers such as barbiturates, carbamazepine, phenytoin, rifampicin; inhibitors such as SSRI antidepressants, cimetidine, diltiazem, macrolides, nitroimidazoles, sedative-hypnotics, verapamil, fluoroquinolones, antihistamines) within four weeks prior to the first dose.; Female participants who have used long-acting estrogen or progestin injections or implants within six months prior to screening; Used any prescription drugs, Chinese herbal medicines, or food supplements (including vitamins, health-care food, etc.) within 2 weeks prior to the first dose; Habitual consumption of grapefruit or grapefruit juice-containing products within 1 week prior to screening, or unwillingness to abstain from grapefruit-containing foods or beverages from 48 hours before dosing of the first period to 48 hours after dosing of the fourth period; Consumption of xanthine-rich foods or beverages (e.g., chocolate, cocoa beans, coffee) within 48 hours prior to the first dose, or unwillingness to abstain from xanthine-rich foods or beverages from 48 hours before the dosing of first period to 48 hours after dosing of the fourth period.

Consumed tea, coffee, and/or foods or beverages containing caffeine within 48 hours prior to the first dose, or do not agree to refrain from consuming tea, coffee, and/or foods or beverages containing caffeine from 48 hours before dosing of the first period until 48 hours after dosing of the fourth period.

* Participants who participated or are participating in any interventional clinical study (including investigational drug or vaccine, and other clinical studies of fluvastatin or other cohorts of this study) and received drugs within 3 months prior to screening.
* Participants with dysphagia or special dietary requirements who cannot adhere to a standardized diet.
* Participants who received live vaccines, attenuated vaccines, or vaccines containing any live viral components within 3 months prior to screening, or those who plan to receive any of these vaccines during the study.
* Participants who experienced blood donation (including component blood donation) or blood loss ≥ 400 mL within 3 months prior to screening; or blood donation (including component blood donation) or blood loss ≥ 200 mL or blood transfusion within 1 month prior to screening; or those who plan to donate blood or blood components during the study or within 1 month after the end of study.
* Participants who experienced major trauma or had a major surgery (e.g., surgery requiring general anesthesia) within 3 months prior to screening, or those who plan to undergo a surgery (except for surgery requiring local anesthesia) during the study or within 3 months after the end of study.
* Participants who have difficulty veins or cannot bear multiple venipunctures, or those with a history of clinically significant fear of needles or hemophobia as judged by the investigator.
* Participants with other diseases or medical history that are clinically significant or may prevent the subjects from completing this study as judged by the investigator (including various systems such as respiratory, cardiovascular, digestive, genitourinary, hematologic, endocrine, neurological, and psychiatric systems, and malignant tumors), or other diseases or medical history that may significantly alter drug absorption, metabolism, or elimination (e.g., history of gastrointestinal surgery, renal surgery, or cholecystectomy, which may affect the in vivo disposition of the drug), or infectious diseases.
* Participants with a history of musculoskeletal and connective tissue disorders (e.g., myalgia, myopathy) or a history of hereditary muscle diseases or rhabdomyolysis.

Participants who are not suitable for participating in this study for any other reasons as judged by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Cmax | up to Day 24
  Observed maximum plasma concentration (Cmax)
AUC0-t | up to Day 24
  Plasma concentration-time curve from time zero extrapolated to the time of last quantifiable concentration (AUC0-t)
AUC0-∞ | up to Day 24
  Plasma concentration-time curve from time zero extrapolated to infinity (AUC0-∞)

CONTACTS AND LOCATIONS:
Overall Officials: Hongying Yang, MD, Principal Investigator — Shenzhen People's Hospital

IPD SHARING:
Plan to Share IPD: No